CLINICAL TRIAL: NCT00111904
Title: Phase II Clinical Trial of Genexol -PM in Patients With Advanced Pancreatic Cancer
Brief Title: Paclitaxel in Treating Patients With Unresectable Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theradex (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000433513; TARGET-S04-10485; WIRB-20050099
Record Dates: First submitted 2005-05-26; First posted 2005-05-27 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2009-06

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; recurrent pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — genexol-PM

INTERVENTIONS:
Drug: paclitaxel-loaded polymeric micelle

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well paclitaxel works in treating patients with unresectable locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the time to progression and time to treatment failure in patients with unresectable locally advanced or metastatic epithelial carcinoma of the pancreas treated with paclitaxel loaded polymeric micelle (Genexol^®-PM).
* Determine the best overall response rate and duration of response in patients treated with this drug.
* Determine the overall survival of patients treated with this drug.
* Determine the clinical benefit and safety of this drug in these patients.

OUTLINE: Patients receive paclitaxel loaded polymeric micelle (Genexol^®-PM) IV over 3 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 43 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed epithelial carcinoma of the pancreas

  * Unresectable* locally advanced or metastatic disease NOTE: *Documented by high-quality contrast-enhanced CT scan
* No known or clinical evidence of CNS metastasis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* SGOT or SGPT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except curatively treated nonmelanoma skin cancer or carcinoma in situ
* No unstable or serious medical condition
* No psychiatric disorder that would preclude giving informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for pancreatic cancer

  * Prior fluorouracil as a radiosensitizer allowed

Endocrine therapy

* Not specified

Radiotherapy

* More than 6 weeks since prior radiotherapy for pancreatic cancer

  * Disease must have progressed after completion of radiotherapy

Surgery

* More than 14 days since prior major surgery and recovered

Other

* More than 30 days since prior investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2005-05; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Time to progression
Time to treatment failure
Best overall response rate
Overall survival
Clinical benefit
Safety

CONTACTS AND LOCATIONS:
Overall Officials: John S. MacDonald, MD, Study Chair — Beth Israel Comprehensive Cancer Center - West Side Campus
Locations (5):
- United States (5):
  - Florida Cancer Specialists - Bonita Springs, Bonita Springs, Florida
  - Midwest Cancer Research Group, Incorporated, Skokie, Illinois
  - Louisiana Oncology Associates - Lafayette, Lafayette, Louisiana
  - St. Vincent's Comprehensive Cancer Center - Manhattan, New York, New York
  - Southwest Regional Cancer Center - Central, Austin, Texas

REFERENCES:
- [Result] Saif MW, Podoltsev NA, Rubin MS, Figueroa JA, Lee MY, Kwon J, Rowen E, Yu J, Kerr RO. Phase II clinical trial of paclitaxel loaded polymeric micelle in patients with advanced pancreatic cancer. Cancer Invest. 2010 Feb;28(2):186-94. doi: 10.3109/07357900903179591. PMID 19968498